CLINICAL TRIAL: NCT02311933
Title: A Randomized Phase II Trial of Tamoxifen Versus Z-Endoxifen HCL in Postmenopausal Women With Metastatic Estrogen Receptor Positive, HER2 Negative Breast Cancer
Brief Title: Tamoxifen Citrate or Z-Endoxifen Hydrochloride in Treating Patients With Locally Advanced or Metastatic, Estrogen Receptor-Positive, HER2-Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-02409; NCI-2014-02409 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A011203; A011203 (Other: Alliance for Clinical Trials in Oncology); A011203 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2014-12-08; First posted 2014-12-09 (Estimated); Results first posted 2021-09-28 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Breast Carcinoma; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (z-endoxifen hydrochloride) (Experimental): Patients receive z-endoxifen hydrochloride PO on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Endoxifen Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm II (tamoxifen citrate) (Experimental): Patients receive tamoxifen citrate PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression and bone metastases may cross over to Arm I and receive z-endoxifen hydrochloride starting no later than 28 days after documentation of disease progression.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Tamoxifen Citrate

INTERVENTIONS:
Drug: Endoxifen Hydrochloride — Given PO
  Other Names: Z-Endoxifen HCl; Z-Endoxifen Hydrochloride
  Arms: Arm I (z-endoxifen hydrochloride)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Tamoxifen Citrate — Given PO
  Other Names: Apo-Tamox; Clonoxifen; Dignotamoxi; Ebefen; Emblon; Estroxyn; Fentamox; Gen-Tamoxifen; Genox; ICI 46,474; ICI 46474; ICI-46474; ICI46474; Jenoxifen; Kessar; Ledertam; Lesporene; Nolgen; Noltam; Nolvadex; Nolvadex-D; Nourytam; Novo-Tamoxifen; Novofen; Noxitem; Oestrifen; Oncotam; PMS-Tamoxifen; Soltamox; TAM; Tamax; Tamaxin; Tamifen; Tamizam; Tamofen; Tamoxasta; Tamoxifeni Citras; Zemide
  Arms: Arm II (tamoxifen citrate)

SUMMARY:
This randomized phase II trial studies how well tamoxifen citrate works compared with z-endoxifen hydrochloride in treating patients with breast cancer that has spread to nearby tissue or lymph nodes or other parts of the body and has estrogen receptors but not human epidermal growth factor receptor 2 (HER2) receptors on the surface of its cells. Estrogen can cause the growth of tumor cells. Hormone therapy using tamoxifen citrate or z-endoxifen hydrochloride may fight breast cancer by lowering the amount of estrogen the body makes. It is not yet known whether tamoxifen citrate or z-endoxifen hydrochloride is more effective in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether progression-free survival with z-endoxifen hydrochloride (HCl) relative to that with tamoxifen (tamoxifen citrate) is prolonged in postmenopausal women with local advanced or metastatic estrogen receptor (ER) positive/Her2 negative breast cancer.

SECONDARY OBJECTIVES:

I. To assess the safety profile of each of these agents in this patient population.

II. To assess whether the tumor response rate (as determined using the Response Evaluation Criteria in Solid Tumors [RECIST] criteria) among those randomized to z-endoxifen HCl differs from that among those randomized to tamoxifen.

III. To estimate the median progression-free survival time for those who receive z-endoxifen HCl after disease progression with tamoxifen.

CORRELATIVE SCIENCE OBJECTIVES:

I. To examine whether ER alpha alterations (defined as either ER activating mutations or ER amplification) are associated with longer progression-free survival (PFS) or higher response rates in the z-endoxifen HCl arm compared to the tamoxifen arm.

II. To determine changes in lipid profiles comparing tamoxifen and z-endoxifen HCl.

III. For each treatment, to evaluate changes in markers of bone formation and absorption after 12 weeks (4 cycles) of treatment.

IV. For all patients and by treatment arm, to determine whether progression-free survival differs with respect to the sensitive to endocrine therapy (SET) index.

V. To examine whether deoxyribonucleic acid (DNA) alterations as measured by Foundation medicine in all coding exons of 287 cancer-related genes as well as 78 polymorphisms in 34 absorption, distribution, metabolism, and excretion (ADME)-related genes are associated with longer PFS or higher response rates in the z-endoxifen HCl arm compared to the tamoxifen arm.

VI. To assess whether the molecular characteristics identified in the tumor biopsies are detectable in the circulating tumor cells (CTCs) and/or cell-free DNA (cfDNA).

VII. For each treatment arm: to examine changes in ER expression on CTCs, changes in estrogen receptor (ESR) mutations or amplification in CTCs or CfDNA and explore the impact of these changes on PFS and response rates.

PHARMACOKINETICS AND PHARMACOGENOMICS OBJECTIVES:

I. To further characterize pharmacokinetics, pharmacogenetics and metabolism of z-endoxifen HCl and tamoxifen.

II. To determine the impact of the concentrations of tamoxifen and its metabolites on PFS in the tamoxifen arm.

III. To determine the impact of the concentrations of z-endoxifen HCl and its metabolites on PFS in the endoxifen arm.

V. To determine the impact of genetic variation in the enzymes responsible for tamoxifen and z-endoxifen HCl metabolism.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive z-endoxifen hydrochloride orally (PO) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive tamoxifen citrate PO once daily (QD) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression and bone metastases may cross over to Arm I and receive z-endoxifen hydrochloride starting no later than 28 days after documentation of disease progression.

After completion of study treatment, patients are followed up yearly for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION ELIGIBILITY CRITERIA
* Women who agree to undergo a standard of care core biopsy of recurrent or metastatic breast cancer to confirm the ER+ (>= 10% nuclear staining) and HER2 negative status
* Patient must have been previously treated with an aromatase inhibitor (either letrozole, anastrozole or exemestane) either in the adjuvant or metastatic setting, and have one of the following types of primary or secondary endocrine resistant disease

  * Primary clinical resistance is defined as one of the following:

    * Recurrence within the first 2 years of adjuvant endocrine therapy while on aromatase inhibitor therapy
    * Progression within first 6 months of initiating first-line endocrine therapy (either aromatase inhibitor or fulvestrant containing regimen) for the treatment of metastatic breast cancer
  * Secondary clinical resistance is defined as one of the following:

    * Recurrence after year 2 while receiving adjuvant aromatase inhibitor therapy, or within 12 months of completing adjuvant aromatase inhibitor therapy
    * Progression occurring 6 or more months after initiating the first endocrine therapy for metastatic disease (either fulvestrant or aromatase inhibitor containing regimen)
* Patients with a history of measurable disease as defined by RECIST criteria or bone only disease are eligible; Note: those patients with non-measurable disease and bone metastases are eligible
* No history of tumors involving spinal cord or heart
* No current evidence of visceral crisis or lymphangitic spread
* No known brain metastases
* Women must be postmenopausal

  * Postmenopausal status is verified by:

    * Prior bilateral surgical oophorectomy, or
    * Age >= 60 years, or
    * Age < 60 with no menses for > 1 year with follicle-stimulating hormone (FSH) and estradiol levels within post menopausal range, according to institutional standard
* Prior treatment

  * No more than two prior chemotherapy regimens in the metastatic setting
  * Prior treatment with an aromatase inhibitor (either anastrozole, letrozole or exemestane), either in the adjuvant or metastatic setting is required
  * Unlimited prior endocrine regimens in the metastatic setting, which may have included an everolimus or cyclin dependent kinase (CDK) 4/6 inhibitor (such as palbociclib, abemaciclib or ribociclib) containing regimen
  * Prior tamoxifen treatment is allowed in the adjuvant setting, but patients must not have experienced relapse within 1 year of stopping tamoxifen
  * No prior treatment with tamoxifen in the metastatic setting
  * No prior treatment with endoxifen
  * Patients who have not fully recovered from acute, reversible effects of prior therapy regardless of interval since last treatment are not eligible to participate in this study

    * EXCEPTION: neuropathies-if grade 2 neuropathies have been stable for at least 3 months since completion of prior treatment patient is eligible
* Not receiving any medications or substances that are strong inhibitors of cytochrome P450 family 2, subfamily D, polypeptide 6 (CYP2D6)
* Not receiving any other investigational agents
* No uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Uncontrolled symptomatic cardiac arrhythmia
  * Uncontrolled hypertension (defined as blood pressure > 160/90)
* None of the following co-morbid conditions:

  * Cataracts of grade 2 or greater as per Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
  * Retinopathy of grade 2 or greater as per CTCAE version 4.0

    * Note: patients that have cataracts that do not require surgery are eligible
    * Note: serious adverse events will be reported on CTEP-Adverse Event Reporting System (AERS) using CTCAE version (v)5.0
  * Deep vein thrombosis/pulmonary embolism (DVT/PE) within the past 6 months

    * Note: patients that are on anticoagulant therapy for maintenance are eligible as long as the DVT and/or PE occurred > 6 months prior to enrollment, and there is no evidence for active thrombosis (either DVT or PE)
* No other active second malignancy other than non-melanoma skin cancers within 3 years of pre-registration; a second malignancy is not considered active if all treatment for that malignancy is completed and the patient has been disease-free for at least 3 years prior to pre-registration
* Eastern Cooperative Oncology Group (ECOG) performance status: 0-2
* Able to swallow oral formulation of the study agent
* Hemoglobin >= 9 g/dL
* Platelet count >= 75,000/mm^3
* Creatinine =< 1.5 x upper limits of normal (ULN)
* Total bilirubin =< 1.5 x upper limits of normal (ULN)
* Aspartate aminotransferase (AST) =< 2.5 x upper limits of normal (ULN); for patients with liver metastasis: =< 5 x upper limits of normal (ULN)
* REGISTRATION ELIGIBILITY CRITERIA
* Patients with either measurable disease as defined by RECIST criteria or bone only disease are eligible; Note: those patients with both non-measurable disease and bone metastases are eligible

  * Non-measurable bone only disease: Non-measurable bone only disease may include any of the following: blastic bone lesions, lytic bone lesions without a measurable soft-tissue component, or mixed lytic-blastic bone lesions without a measurable soft-tissue component
  * Lytic bone lesions, with an identifiable soft tissue component, evaluated by computed tomography (CT) or magnetic resonance imaging (MRI), can be considered as measurable lesions if the soft tissue component otherwise meets the definition of measurability previously described
* No tumors involving spinal cord or heart
* No visceral crisis, lymphangitic spread or known brain metastases: visceral crisis is not the mere presence of visceral metastases, but implies severe organ dysfunction as assessed by symptoms and signs, laboratory studies, and rapid progression of disease
* Histologic confirmation, from the A011203 pre-registration biopsy, by institutional/local pathologist of either locally advanced or metastatic breast cancer that is estrogen receptor positive and HER2 negative; those patients with bone only disease with either no tumor or insufficient tumor for ER/progesterone receptor (PR) and HER2 staining after the bone biopsy are still eligible to participate in this study
* Estrogen receptor positive disease is defined as > 10% nuclear staining
* HER2 negative disease as per 2013 American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines, one of the following must apply:

  * 0 or 1+ by immunohistochemistry (IHC) and not amplified by in situ hybridization (ISH)
  * 0 or 1+ by IHC and ISH not done
  * 2+ by IHC and not amplified by ISH or
  * IHC not done and not amplified by ISH
* None of the following therapies are allowed prior to registration:

  * Chemotherapy =< 2 weeks
  * Immunotherapy =< 2 weeks
  * Biologic therapy =< 2 weeks
  * Hormonal therapy =< 2 weeks
  * Monoclonal antibodies =< 2 weeks
  * Radiation therapy =< 2 weeks
  * Anti-Her-2 or other "targeted" (e.g. mammalian target of rapamycin [mTOR]) therapy =< 2 weeks

    * NOTE : Any toxicities derived from these therapies must be =< grade 2 prior to starting study therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2026-02-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Goetz, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (561):
- United States (561):
  - Southern Cancer Center PC-Providence, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mercy Cancer Center, Merced, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center - Saint Joseph Hospital, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Ascension Alexian Brothers - Elk Grove Village, Elk Grove Village, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - JCHC McCreery Cancer Center, Fairfield, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Gaston Hematology and Oncology Associates-Belmont, Belmont, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Gaston Hematology and Oncology Associates, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Maria Parham Hospital, Henderson, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Scotland Memorial Hospital-Laurinburg Cancer Center, Laurinburg, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Cleveland Hematology and Oncology Associates PC, Shelby, North Carolina
  - Johnston Memorial Hospital, Smithfield, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Z-endoxifen Hydrochloride): Patients receive 80 mg z-endoxifen hydrochloride PO on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Arm II (Tamoxifen Citrate): Patients receive 20 mg tamoxifen citrate PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression and bone metastases may cross over to Arm I and receive z-endoxifen hydrochloride starting no later than 28 days after documentation of disease progression.
Period: Overall Study
Arm/Group | Arm I (Z-endoxifen Hydrochloride) | Arm II (Tamoxifen Citrate)
Started | 41 | 40
Completed | 41 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients registered were included in the baseline characteristics analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Z-endoxifen Hydrochloride) | Arm II (Tamoxifen Citrate) | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Continuous [Median (Full Range); unit: years] | 64 [48 to 83] | 66 [46 to 80] | 65 [46 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 40 | 81
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 39 | 36 | 75
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 36 | 36 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: The primary endpoint is progression-free survival (PFS) defined as the time from randomization to documentation of local, regional or distant disease progression or death without progression of disease.
Time Frame: Assessed up to 5 years
Population: All patients registered who began protocol treatment and were eligible for assessment were included in this analysis. One patient in Arm I was ineligible, two patients in Arm II were ineligible and one patient in Arm II did not receive treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm I (Z-endoxifen Hydrochloride) | Arm II (Tamoxifen Citrate)
Number analyzed (Participants) | 40 | 37
days | 130 [76 to 138] | 42 [24 to 129]

2. Secondary Outcome: Incidence of Adverse Events, Per Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: For a given adverse event (AE), the proportion of patients on each treatment arm who report developing a grade 2-5 of this AE will be determined.
Time Frame: Up to 5 years
Reporting Status: Not Posted

3. Secondary Outcome: Tumor Response Rate by Study Arm, Defined as the Number of Patients With a Complete or Partial Response
Description: Defined by Response Evaluation Criteria in Solid Tumors on 2 consecutive evaluations at least 6 weeks apart, divided by the total number of eligible patients who began study treatment. A 90% binomial confidence interval will be constructed for the true response rate.
Time Frame: Up to 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival Distribution by Study Arm
Description: The distribution of survival times will be estimated using the method of Kaplan-Meier.
Time Frame: The time from registration to death due to any cause, assessed up to 5 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Deoxyribonucleic Acid (DNA) Alterations as Measured by Foundation Medicine
Description: Data will be returned as presence or absence of various DNA alterations, along with description of type and location of the alteration. The nature of alterations in each pathway and gene will be described in tabular format. Association of presence or absence of DNA alterations with PFS will be assessed overall, by pathway, and by gene via Cox regression with the goal of evaluating hazard ratio estimates and confidence intervals. Alterations will be considered together as well as by type. Model fit and stability evaluated, and exact methods used if needed. Performed for both arms and within arms.
Time Frame: Baseline
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Nuclear Receptor Coactivator 3 (SRC3) Immunohistochemistry Expression Levels
Description: Within each treatment arm, a point and interval estimate of the difference in tumor response rate between those with metastatic SRC3-positive disease and those with metastatic SRC3-negative disease will be constructed using the properties of the binomial distribution. Also, a point and interval estimate of the odds of disease progression among those with metastatic SRC3-positive disease relative to those with metastatic SRC3-negative disease will be ascertained from the parameter estimates of fitting a proportional hazard model to the progression data.
Time Frame: Baseline
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Biochemical Markers of Bone Turnover
Description: For each of the markers of bone formation, the percent change after 2 courses of treatment from pre-treatment levels will be determined. A two-sided alpha = 0.01 z-test will be used to assess whether the percent change in a given bone absorption biomarkers differs with respect to treatment.
Time Frame: Baseline to week 8 (after course 2)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Z-endoxifen Hydrochloride Area Under Curve (AUC)
Description: A population PK will be developed using the software program NONMEM, Version 7. The model will be parameterized in terms of AUC (the primary endpoint), as well as clearance and volume of distribution. Criteria for model selection will include the likelihood ratio test, shrinkage estimates, reasonableness of parameter estimates, as well as goodness-of-fit plots. Attempts will be made to identify the covariates that affect drug behavior or those that explain variability in this patient population.
Time Frame: Baseline, 2-4, and 4-6 hours post-administration day 1 of course 1; baseline day 2 of course 1; pre-administration day 1 of course 3; pre-administration day 1 of course 9
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Pharmacokinetic (PK) Data
Description: Examined in an exploratory and hypothesis-generating fashion. Pharmacokinetic-pharmacodynamic (PD) relationships will be explored for effects of endoxifen on efficacy-related, adverse events or laboratory parameters of clinical interest. Exploratory/graphical analyses will be conducted for PK/PD evaluations and may be followed by model-based analyses. The data may be pooled with data from other/future studies for additional population PK/PD analyses.
Time Frame: as for outcome 8
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Pharmacogenetic Data
Description: Examined in an exploratory and hypothesis-generating fashion.
Time Frame: Baseline
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Pharmacodynamic Data
Description: PK/PD relationships will be explored for effects of endoxifen on efficacy-related, adverse events or laboratory parameters of clinical interest. Exploratory/graphical analyses will be conducted for PK/PD evaluations and may be followed by model-based analyses. The data may be pooled with data from other/future studies for additional population PK/PD analyses.
Time Frame: as for outcome 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected at the end of every 3 week cycle (up to a max 92 cycles). The data reported here for the primary submission is through 8/18/2021.
Description: Adverse events were collected at the end of every 3 week cycle (up to a max 92 cycles). The data reported here for the primary submission is through 8/18/2021.
Arm/Group | Arm I (Z-endoxifen Hydrochloride) | Arm II (Tamoxifen Citrate)
All-Cause Mortality (participants affected / at risk) | 1/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 8/41 | 11/39
Other Adverse Events (participants affected / at risk) | 34/41 | 36/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Z-endoxifen Hydrochloride) (N=41) | Arm II (Tamoxifen Citrate) (N=39)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Z-endoxifen Hydrochloride) (N=41) | Arm II (Tamoxifen Citrate) (N=39)
Anemia (Blood and lymphatic system disorders) | 5 (6) | 4 (20)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 0 (0) | 1 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Blurred vision (Eye disorders) | 0 (0) | 2 (8)
Dry eye (Eye disorders) | 0 (0) | 1 (4)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (8)
Constipation (Gastrointestinal disorders) | 6 (13) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (7) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (23) | 3 (8)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (4)
Nausea (Gastrointestinal disorders) | 5 (10) | 7 (11)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 2 (6) | 0 (0)
Fatigue (General disorders) | 16 (57) | 7 (48)
Fever (General disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 2 (2) | 1 (2)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (5) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (2) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 3 (6)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Vulval infection (Infections and infestations) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Alkaline phosphatase increased (Investigations) | 3 (11) | 3 (10)
Aspartate aminotransferase increased (Investigations) | 9 (26) | 14 (57)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (2)
Cholesterol high (Investigations) | 2 (7) | 2 (4)
Creatinine increased (Investigations) | 2 (4) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (24) | 3 (5)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (6)
Platelet count decreased (Investigations) | 2 (2) | 3 (4)
Weight loss (Investigations) | 1 (4) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 2 (8)
Anorexia (Metabolism and nutrition disorders) | 7 (24) | 3 (7)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (14) | 4 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 2 (4)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 16 (61) | 13 (84)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (11) | 4 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 4 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 3 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (10) | 1 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (8)
Dizziness (Nervous system disorders) | 2 (4) | 2 (6)
Dysgeusia (Nervous system disorders) | 3 (16) | 2 (23)
Headache (Nervous system disorders) | 1 (2) | 3 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (7) | 0 (0)
Spasticity (Nervous system disorders) | 0 (0) | 1 (2)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 5 (24)
Irritability (Psychiatric disorders) | 0 (0) | 1 (4)
Urinary frequency (Renal and urinary disorders) | 1 (4) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (7)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (2) | 1 (2)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 4 (30)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 1 (5)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (7)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (6) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 0 (0) | 1 (2)
Hot flashes (Vascular disorders) | 25 (115) | 20 (178)
Hypertension (Vascular disorders) | 2 (10) | 4 (8)
Thromboembolic event (Vascular disorders) | 1 (4) | 3 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT02311933/Prot_SAP_000.pdf